CLINICAL TRIAL: NCT06000878
Title: Evaluate the Effectiveness of First Aid E-book Intervention on First Aid Knowledge, Self-efficacy, and Skills Among New Nurses
Brief Title: Evaluate the Effectiveness of First Aid E-book Intervention Among New Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KMUHIRB-SV(I)-20210025
Record Dates: First submitted 2023-07-14; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2022-01

CONDITIONS: First Aid; Knowledge; Self-efficacy
Keywords: e-book; first aid knowledge; self-efficacy; first aid skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The experimental group received a one-hour e-book course plus one month of first aid e-book intervention and regular training
  Interventions: Other: first aid e-book
- control group (No Intervention): The control group only received one month of regular training.

INTERVENTIONS:
Other: first aid e-book — interactive first aid e-book interventions
  Arms: experimental group

SUMMARY:
Background: First aid skills are clinical performance ability requiring a higher level of skills for new nurses. At present, the focus of first aid-related teaching materials and methods remain on books and physical courses. E-books have not yet been applied to first aid skills training for new nurses despite their advantage of making reading, learning, and reviewing available at any time.

Objective: To assess the effect of receiving interactive first aid e-book interventions on new nurses in a medical center in southern Taiwan in respect of first aid knowledge, self-efficacy, and first aid skills.

Methods: A two-group three-time repeated measures experimental design was adopted. 70 qualified new nurses were randomly assigned to the experimental group and the control group, each composed of 35 nurses. The experimental group received a one-hour e-book course plus one month of first aid e-book intervention and regular training, whereas the control group only received one month of regular training. Performance indicators included administering the objective structured clinical examination (OSCE) on first aid skills, and questionnaires for knowledge and self-efficacy related to first aid skills. The experimental group received qualitative interviews and filled out the system usability scale one month after the intervention. Data were analyzed using the independent samples t-test, chi-squared test, paired samples t-test, and generalized estimating equations (GEE).

DETAILED DESCRIPTION:
1. Introduction Paramedics are the first-line medical personnel on the emergency scene and can help in effectively treating the medical condition in the first few minutes. For instance, Cardiopulmonary resuscitation (CPR) can improve the chances of survival of cardiac arrest patients (Partiprajak & Thongpo, 2016 ; P. Y. Hsieh et al., 2021). CPR is an attempt to restore spontaneous circulation through chest compressions when the patient is not breathing and the heart is beating (Suseel et al., 2019). Crucially, the ability to perform effective CPR immediately requires repeated first aid training (Roh & Issenberg, 2014 ; Moon & Hyun, 2019). However, among clinical skills, new nurses find it most difficult to perform CPR (Liou et al., 2020). If new recruits lack professional training or confidence in their abilities, the quality of first aid provided by them may be affected (Ihunanya et al., 2020). Therefore, it is imperative to implement a well-designed training program that effectively equips clinical nurses with the necessary first aid knowledge and skills. (P. Y. Hsieh et al., 2021).
2. Method 2.1 Design and participants This study used an experimental two-group pre- and post-test design. Three repeated measures were taken: pre-test (T0), immediate post-test (T1), and one-month post-test (T2). The one-month post-test was used to detect new nursing care personnel's retention of first aid knowledge, self-efficacy, and first aid skills. G power 3.1.9.2 version was used to estimate the number of samples using repeated measures ANOVA. The effect size was set to 0.3 (Kotrlik & Williams, 2003), alpha value was set to 0.05, detection power was 0.8, and correlation value was 0.5. The measurement was repeated thrice. As such, the total number of samples required should be 62 bits. Considering an estimated attrition rate of 10% or 7 people, the total number of cases accepted was 70. The main investigator explained the purpose and process of the study to the new nurses in each ward and invited them to participate in the study. Data was collected between August 2021 and October 2021. The sample inclusion criteria were that participants were newly recruited nurses within two years with a basic first aid BLS certificate. Meanwhile, those who were unable to perform CPR due to hand injuries were excluded. A computer was used to randomly assign the 70 eligible new nurses in the medical center to the experimental and control groups, with 35 each.

2.2 Study protocol The experimental group took a one-hour e-book course plus one month of first aid e-book intervention and routine training, whereas the control group received only one month of routine training. Effectiveness indicators were measured at pre-test (T0), immediate post-test (T1), and one-month post-test (T2). In order to assess the effectiveness of the first aid e-book intervention, the first aid skill Objective Structured Clinical Examination (OSCE) evaluation form was utilized alongside self-efficacy questionnaires for first aid knowledge and first aid ability. This comprehensive approach aimed to evaluate the effectiveness of the intervention.

2.3 Research tool The research tools included the basic demographic data sheet, first aid knowledge questionnaire, first aid self-efficacy scale, first aid skills OSCE evaluation form, and system usability scale (SUS).

2.3.1 Demographic basic data sheet The demographic basic data sheet was exclusively utilized during the pre-test (T0) phase. It encompassed details such as gender, age, education level, clinical experience, previous participation in first aid training courses, and the number of times the participants had engaged in first aid activities.

2.3.2 First aid knowledge questionnaire The first aid knowledge questionnaire was based on the 2020 American Heart Association First Aid Guidelines Update (Cummins & Hazinski, 2020), and American Heart Association Cardiopulmonary Resuscitation and Cardiovascular Emergency Guidelines (Craig-Brangan & Day, 2020). The questionnaire included five items with a total of 20 questions to test the new nurses' concept and understanding of first aid: first aid assessment and initial treatment (four questions), maintenance of airway and circulation (four questions), interpretation and treatment of abnormal heart rhythm (five questions), teamwork and abnormal handling (six questions), and communication and coordination with the patient's family members (one question). Each question is 5 points and measured on a five-point scale, with the total score being 0 to 100 points for 20 questions. The higher the score, the better was the awareness of first aid. The self-made first aid knowledge questionnaire, assessed by three experts, demonstrated a Content Validity Index (CVI) of 0.93, indicating a high level of content validity. The Cronbach's α value of the internal consistency reliability of the scale was 0.713, indicating an acceptable level of internal consistency.

2.3.3 First aid self-efficacy scale This study modified the "Self-efficacy Scale of First Aid Ability for Nurses" developed by Xie et al. (2014) to measure the self-efficacy of first aid ability assessed by new nurses themselves (Xie et al., 2014). The self-efficacy scale has six items with a total of 30 questions: maintenance of the respiratory tract and circulation (seven questions), teamwork and abnormal handling (twelve questions), communication and coordination between patients and their families (three questions), and abnormal heart rhythm interpretation and treatment (three questions), first aid assessment and initial treatment (four questions), demonstration of nursing first aid role and function (one question). Each question was answered on a five-point Likert Scale, with a total score ranging between 30-150 points; the higher the score, the higher the confidence level. The modified first aid self-efficacy scale demonstrated a content-related validity CVI value of 0.94, indicating strong expert agreement on the content relevance. Furthermore, the internal consistency reliability of the scale, measured by Cronbach's α value, was 0.964, signifying excellent internal consistency.

2.3.4 First aid skills OSCE A modified first aid skill measurement OSCE based on Li Huizhen et al. (2016) OSCE was used (Li Huizhen et al., 2016). A standardized clinical scenario was employed, and the examiner provided prompts during the test to assess the participants' first aid skills. The test was divided into three dimensions, with a total of 30 questions. The first dimension was pre-emergency assessment, performing cardiac compressions, and first aid balls (9 questions). The second dimension was the use of electric shock device and electric shock, and placing the endotracheal tube to confirm the position and fix it (11 questions). The third dimension was communication and coordination between first aid administration, and patient's family members (10 questions). The test time was 15 min, and each question was scored on five points. The total score on this scale ranges from 0 to 150 points. The higher the score, the better the first aid skill. Here, the CVI value of the OSCE evaluation form was 0.97 and Cronbach's α value of the internal consistency reliability of the scale was 0.964, indicating strong the expert content-related validity and excellent internal consistency .

2.3.5 First aid e-book The interactive first aid e-book was produced by SimMAGIC eBook, an interactive multimedia e-book editing software developed by Hama Star Technology. The interactive functions of the e-book included clicking, covering, dragging, scratching, linking, preset questions, and timely feedback. For each first aid concept, we provided multimedia learning materials, such as pictures and video explanations. Individuals can click "Play" and watch videos. The content of the e-book includes basic first aid knowledge and first aid drug knowledge, basic cardiopulmonary resuscitation first aid skills, assisting intubation, electric shock device operation video, how to perform team first aid practical operation teaching video, and interpretation and treatment of fatal arrhythmia. At the end, we designed some first aid concept knowledge about self-assessment, with interactive operation questions and answers to increase learning interest and enhance learning motivation. Then, we uploaded the e-book to the website and linked the URL into a QR code so that new nursing staff could use mobile phones, tablets, or computers to learn.

2.3.6 System usability scale (SUS) John Brooke constructed the SUS in 1986. SUS has been used to measure various products, system interfaces, and services, including websites, mobile phones, and applications. It has 10 items which are measured on a five-point Likert scale from 1 = strongly disagree to 5 = strongly agree. Questions 1, 3, 5, 7, and 9 were positive questions, and questions 2, 4, 6, 8, and 10 were negative questions. The calculation method was as follows: subtract 1 from the score of the positive question, subtract the score of each question from 5 for the negative question, add up the scores of all questions, and multiply by 2.5 to get the average score of system usability (Wang et al., 2020). The SUS score was divided into six grades to represent the overall usability of the product: 90-100 were labelled A grade, representing super easy to use (best imaginable); 80-89 were labelled B grade, representing excellent use (excellent); 70-79 were labelled C Grade, representing good (good), grades 60-69 represent D-grades (ok), and grades 0-59 represent F-grades (poor) (Bangor, 2009). The CVI value of the expert content-related validity of the modified system usability scale is 0.90.

2.3.7 Qualitative interview Finally, interviews were conducted with participants in a confidential discussion room. The interviews were recorded and the content was kept confidential to ensure the reliability and authenticity of the data collection. Six new nurses were interviewed, who had become nurses in the past two years and had just completed the second post-test of the e-book intervention. The outline of the interview was structured on the following questions: 1. How helpful do you think the first aid e-book is? 2. What devices do you use to read e-books? 3. What do you think about the first aid e-book compared with other BLS courses? Which one do you prefer? Why? This study adopted the data analysis method of Colaizzi (1978). Specifically, We performed a systematic analysis, induction, and translation, categorizing the shared characteristics of these meanings into distinct themes.

ELIGIBILITY:
Inclusion Criteria:

* In medicine within 2 years after graduation New nurses working in the center who have passed the probationary period and have a basic first aid BLS certificate.
* Willing to participate with this researcher.

Exclusion Criteria:

* Injured hands and unable to perform CPR

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
First Aid Knowledge Questionnaire | pre-test, immediate post-test, and one-month post-test
  The first aid knowledge questionnaire was based on the 2020 American Heart Association First Aid Guidelines Update (Cummins & Hazinski, 2020), and American Heart Association Cardiopulmonary Resuscitation and Cardiovascular Emergency Guidelines (Craig-Brangan & Day, 2020). The questionnaire included five items with a total of 20 questions to test the new nurses' concept and understanding of first aid: first aid assessment and initial treatment (four questions), maintenance of airway and circulation (four questions), interpretation and treatment of abnormal heart rhythm (five questions), teamwork and abnormal handling (six questions), and communication and coordination with the patient's family members (one question). Each question is 5 points and measured on a five-point scale, with the total score being 0 to 100 points for 20 questions. The higher the score, the better was the awareness of first aid.
First Aid Self-Efficacy Scale | pre-test, immediate post-test, and one-month post-test
  This study modified the "Self-efficacy Scale of First Aid Ability for Nurses" developed by Xie et al. (2014) to measure the self-efficacy of first aid ability assessed by new nurses themselves (Xie et al., 2014). The self-efficacy scale has six items with a total of 30 questions: maintenance of the respiratory tract and circulation (seven questions), teamwork and abnormal handling (twelve questions), communication and coordination between patients and their families (three questions), and abnormal heart rhythm interpretation and treatment (three questions), first aid assessment and initial treatment (four questions), demonstration of nursing first aid role and function (one question). Each question was answered on a five-point Likert Scale, with a total score ranging between 30-150 points; the higher the score, the higher the confidence level.
First aid skills OSCE | pre-test, immediate post-test, and one-month post-test
  A modified first aid skill measurement OSCE based on Li Huizhen et al. (2016) OSCE was used (Li Huizhen et al., 2016). A standardized clinical scenario was employed, and the examiner provided prompts during the test to assess the participants' first aid skills. The test was divided into three dimensions, with a total of 30 questions. The first dimension was pre-emergency assessment, performing cardiac compressions, and first aid balls (9 questions). The second dimension was the use of electric shock device and electric shock, and placing the endotracheal tube to confirm the position and fix it (11 questions). The third dimension was communication and coordination between first aid administration, and patient's family members (10 questions). The test time was 15 min, and each question was scored on five points. The total score on this scale ranges from 0 to 150 points. The higher the score, the better the first aid skill.

SECONDARY OUTCOMES:
System usability scale (SUS) | one-month post-test
  SUS has been used to measure various products, including websites, mobile phones, and applications (John Brooke, 1986). It has 10 items which are measured on a five-point Likert scale from 1 to 5. Questions 1, 3, 5, 7, and 9 were positive questions, and questions 2, 4, 6, 8, and 10 were negative questions. The calculation method was as follows: subtract 1 from the score of the positive question, subtract the score of each question from 5 for the negative question, add up the scores of all questions, and multiply by 2.5 to get the average score of system usability (Wang et al., 2020). The SUS score was divided into six grades to represent the overall usability of the product: 90-100 were labelled A grade, representing super easy to use (best imaginable); 80-89 were labelled B grade, representing excellent use (excellent); 70-79 were labelled C Grade, representing good (good), grades 60-69 represent D-grades (ok), and grades 0-59 represent F-grades (poor) (Bangor, 2009).
Qualitative interview | one-month post-test
  1. How helpful do you think the first aid e-book is? 2. What devices do you use to read e-books? 3. What do you think about the first aid e-book compared with other BLS courses? Which one do you prefer? Why?

CONTACTS AND LOCATIONS:
Overall Officials: CHIA-KUEI HU, Study Director — Kaohsiung Medical University Hospital, Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung Medical University, Kaohsiung City, No.100, Tzyou 1st Rd., Sanmin District, Taiwan

IPD SHARING:
Plan to Share IPD: No